CLINICAL TRIAL: NCT05433974
Title: Pre-therapeutic Analysis of the Individual Radiosensitivity of Cancer Patients in Luxembourg (APRI-Lux): Prospective National Interventional Study With Minimal Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Francois Baclesse, Luxembourg (Other)
Collaborators: BIONEXT (Unknown); Neolys (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: APRI-Lux
Record Dates: First submitted 2022-06-20; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Radiosensitivity; Cancer; Radiation Toxicity
MeSH Terms: conditions — Neoplasms; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiosensitivity (Other): Patient who agree to participate in this research study will have blood sample collected in order to perform the RadioDtect test.
  Interventions: Biological: Blood sample collection

INTERVENTIONS:
Biological: Blood sample collection — Blood sample collection : 2 X 6 mL

SUMMARY:
Pre-therapeutic analysis of the individual radiosensitivity of cancer patients in Luxembourg

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient with an indication for curative radiotherapy
* Patient having given his signed written informed consent before any specific procedure of the protocol.

Exclusion Criteria:

* Patient with a contraindication to radiotherapy
* Patient with an indication for palliative radiotherapy
* Patient with a history of radiotherapy in the area where the cancer is located
* Patient unable to submit to the medical follow-up of the trial for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Validation of RadioDtect test on early radiation-induced toxicity | 3 months
  prospectively validate the predictive capacities of the RadioDtect individual radiosensitivity blood test on early radiation-induced toxicity. The validation will be based on ATM protein assay and rate of acute toxicities of grade ≥ 2 to 3 months according to NCI-CTCAE v4.03 criteria

SECONDARY OUTCOMES:
Validation of RadioDtect test on delayed radiation-induced toxicity | 12 months
  to prospectively validate the predictive capacities of the RadioDtect individual. radiosensitivity blood test on delayed radiation-induced toxicity at 12 months. The validation will be based on ATM protein assay and rate of acute toxicities of grade ≥ 2 to 3 months according to NCI-CTCAE v4.03 criteria

IPD SHARING:
Plan to Share IPD: Undecided